CLINICAL TRIAL: NCT04380662
Title: RRisk Factors Worsening COVID19 (Coronavirus Infectious Disease 2019) for Outpatient With Home Monitoring (COVID-A-DOMEVA Study)
Brief Title: Risk Factors Worsening COVID19 for Out-patient With Home Monitoring
Acronym: COVIDADOMEVA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.135; 2020-A01040-39 (Other: ID RCB)
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Covid19
Keywords: RISK FACTOR; HEALTH STATUS; CLINICAL CARE PATHWAY; COVID19; COHORT; OUT PATIENT
MeSH Terms: conditions — COVID-19 | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID+ patients WITH worsening of the disease: COVID+ patients WITH worsening of the disease (case group)
  Interventions: Other: Risk factors
- COVID+ patients WITHOUT worsening of the disease: COVID+ patients WITHOUT worsening of the disease (control group)

INTERVENTIONS:
Other: Risk factors — The studied potential risk factors will be the following:
  * Socio-demographic: age, sex, place of residence, CSP and income.
  * Comorbidities or aggravation: COPD, asthma, immunosuppression, or heart failure, diabetes imbalance, etc.
  * Clinical signs: asthenia, dyspnea (kinetics), blood sugar, nutritional status, weight gain…
  * Drugs other than those related to the infection and potential self-medication (anti-inflammatory, CEI, ARA…)
  Groups: COVID+ patients WITH worsening of the disease

SUMMARY:
The main objective of the COVIDADOMEVA study is to identify the risk factors aggravating the COVID-19 (risk or protective factors), in out-patients suspected of being infected with precocious home monitoring.

The primary event defining the aggravation will be then: hospitalization (medicine, resuscitation) or death.

The studied potential risk factors will be mainly:

* Socio-demographic: age, sex, place of residence or income
* Comorbidities
* Clinical signs: asthenia, dyspnea (kinetics)…
* Drugs other than those related to the infection

For this research project, this study needs to use the patient's data of the COVIDADOM cohort (patients suspected of being infected with SARS-CoV-2 with home monitoring) and will collect some supplementary data (clinical and biological). All these data will be integrated and analyzed in the PREDIMED clinical data lake platform (The implementation of PREDIMED has been approved by the French authority in terms of GDPR, CNIL, on October 10, 2019).

DETAILED DESCRIPTION:
In front of the recent emergence of the SARS-CoV-2 coronavirus (COVID) in December 2019 in the Wuhan region of China, knowledge of the clinical course and of the aggravating risk factors linked to this virus is still incomplete.

COVID is associated with severe morbidity and an estimated mortality of 2-4% in patients without comorbidity. According to a WHO report published on the situation in China, patients with serious chronic pathologies, such as diabetes or severe obesity, are particularly vulnerable and mortality rates were higher: from 7 to 13%.

Monitoring and describing the clinical pathway of out-patients suspected of being infected according to their medical history should improve knowledge of COVID, and then adapt patient care management and control the COVID pandemic.

Currently, few European studies have described the potential risk factors that could lead to the worsening of the disease. Since the March 16th, the university hospital of Grenoble (France) has developed an information technology system to monitor out-patients suspected of being infected with SARS-CoV-2 coronavirus and with early home monitoring: the COVIDADOM cohort

That's why the COVIDADOMEVA study is then to identify the risk factors aggravating the COVID, in out-patients with precocious home monitoring.

The primary event defining the aggravation will be then: hospitalization (medicine, resuscitation) or death

The studied potential risk factors will be the following:

* Socio-demographic: age, sex, place of residence, CSP, and income.
* Comorbidities or aggravation: COPD, asthma, immunosuppression, or heart failure, diabetes imbalance, etc.
* Clinical signs: asthenia, dyspnea (kinetics), blood sugar, nutritional status, weight gain…
* Drugs other than those related to the infection and potential self-medication (anti-inflammatory, CEI, ARA…)

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical symptomatology suspecting COVID-19, that is to say: severe dyspnea, and/or serious extra pulmonary signs (myalgia, diarrhea, etc.) OR
* Patient with clinical symptomatology (cough or dyspnea or fever with ENT signs) AND at least one of the following comorbidities: COPD stage 1 or 2 (dyspnea usually absent or for marked efforts), Asthma with daily inhaled corticosteroid therapy, Immunosuppression or cancer during chemotherapy, Coronary history, Heart failure (Stages 2 and 3, dyspnea with moderate or low effort), Obesity (BMI> 30), Type 1 or 2 diabetes, cirrhosis from Child B, pregnant woman in the 3rd trimester.
* Patient with a phone monitoring of at least more than 2 calls, if no aggravation of disease.

Exclusion Criteria:

* Person deprived of liberty by judicial or administrative decision
* Person being subject to a legal protection measure
* Person who expressed opposition to participating in the COVIDADOMEVA study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients included in the study are from the Grenoble area, had contacted the accident and emergency ward (A&E department) or their general practitioner (GP). The patients recruited are patients suspected of being infected with SARS-CoV-2, with home monitoring including the containment measures set up according to the French Health recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Identify the factors associated with the worsening of the COVID19 | 30 days
  The event defining the aggravation will be: hospitalization (medicine, resuscitation) or death
  The main potential risk factors will be the following:
  * Socio-demographic: age, sex, place of residence, CSP and income.
  * Comorbidities or aggravation: COPD, asthma, immunosuppression, or heart failure, diabetes imbalance, etc.
  * Clinical signs: asthenia, dyspnea (kinetics), blood sugar, nutritional status, weight gain…
  * Drugs other than those related to the infection and potential self-medication (anti-inflammatory, CEI, ARA…)

SECONDARY OUTCOMES:
Describe the clinical care pathway of patients from Day 0 to Day 14 | 30 days
  Clinical and monitoring data of the the COVIDADOM cohort and of the COVIDADOMEVA case report form (CRF)
Describe the health status at Day 30 | 30 days
  Health status patient (stay at home, hospitalization or death)
Describe the quality of life during the disease | 30 days
  EQ5D-5L score

CONTACTS AND LOCATIONS:
Overall Officials: Olivier EPAULARD, MD-PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Fang L, Karakiulakis G, Roth M. Are patients with hypertension and diabetes mellitus at increased risk for COVID-19 infection? Lancet Respir Med. 2020 Apr;8(4):e21. doi: 10.1016/S2213-2600(20)30116-8. Epub 2020 Mar 11. No abstract available. PMID 32171062
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] OMS. Soins à domicile pour les patients COVID-19 qui présentent des symptômes bénins, et prise en charge de leurs contacts. Lignes directrices provisoires, 17 mars 2020 (5pages). WHO reference number : WHO/2019-nCoV/IPC/HomeCare/2020.3
- [Background] Jordan RE, Adab P, Cheng KK. Covid-19: risk factors for severe disease and death. BMJ. 2020 Mar 26;368:m1198. doi: 10.1136/bmj.m1198. No abstract available. PMID 32217618